CLINICAL TRIAL: NCT04062110
Title: Below-elbow or Above-elbow Cast for Conservative Treatment of Extra-articular Distal Radius Fractures With Dorsal Displacement: a Prospective Randomized Trial
Brief Title: Below-elbow or Above-elbow Cast for Extra-articular Distal Radius Fractures
Acronym: UNIFE/GC01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 161184
Record Dates: First submitted 2019-06-21; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-06

CONDITIONS: Radius Fractures
Keywords: distal radius fractures; above-elbow cast; below-elbow cast; conservative treatment; extra-articular fractures
MeSH Terms: conditions — Radius Fractures; Wrist Fractures | interventions — Casts, Surgical

STUDY DESIGN:
Intervention Model Description: two-arm, parallel-group, prospective randomised trial
Who Masked: Participant
Masking Description: randomised trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long plaster casts for type AO 2R3A2.2 (Active Comparator): Closed reduction of the fracture and immobilization with long plaster casts (above-elbow, Long plaster casts).
  Interventions: Device: plaster cast
- Short plaster casts for type AO 2R3A2.2 (Active Comparator): Closed reduction of the fracture and immobilization with short plaster casts (below-elbow, Short plaster casts)
  Interventions: Device: plaster cast

INTERVENTIONS:
Device: plaster cast — Closed Reduction of Fracture and Application of Plaster Cast

SUMMARY:
The aim of this prospective randomised study was to shed more light on the issue by comparing the capacity of long plaster casts (above-elbow, LC) and short plaster casts (below-elbow, SC) to maintain the reduction of extra-articular distal radius fractures with dorsal displacement (2R3A2.2, according to the AO/OTA classification). The initial hypothesis was that the short cast would be equally as effective as the long cast in treating this type of fracture. The secondary objective of the study was to determine whether or not there is a direct correlation between radiological parameters and functional outcomes in such patients.

DETAILED DESCRIPTION:
Distal radial fractures are common traumatic injuries, but their management remains controversial, Hence, we conducted a two-arm, parallel-group, prospective randomised trial to compare the capacity of long casts (above-elbow) and short casts (below-elbow) to maintain the reduction of extra-articular distal radius fractures with dorsal displacement (AO/OTA classification: 2R3A2.2). Eligible patients with AO/OTA 2R3A2.2 fractures treated with closed reduction and cast immobilization were randomized to the long cast group or to the short cast group. Baseline radiological parameters, radial inclination (RI), radial height (RH), ulnar variance (UV) and palmar tilt (PT) were taken, and compared with clinical (DASH, Mayo Wrist and Mayo Elbow) and radiological scores taken at 7-10 days, 4 weeks and 12 weeks. Furthermore, to evaluate correlations between radiological parameters and functional outcomes, patients were divided into two groups according to whether or not their radiological parameters at Follow-ups 2 and 3 were acceptable, i.e. within the range 11-12 mm for RH, 16°-28° for IR, -4-+2 mm for UV, and 0°-22° for PT.

ELIGIBILITY:
Inclusion Criteria:

* extra-articular fractures of the distal radius with dorsal displacement (type 2R3A2.2 according to the AO classification).
* eligible for conservative treatment with plaster

Exclusion Criteria:

* open fractures
* extra-articular distal radius fracture with volar displacement
* a history of allergy to the cast material
* patients scheduled for surgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
To measure the maintenance of fracture reduction according to radial inclination (Long plaster casts Vs Short plaster casts) | compared at baseline, at 7-10 days, at 4 weeks and at 12 weeks
  Radial inclination: angle of the distal radial surface with respect to a line perpendicular to the shaft, a normal 16° - 18°
To measure the maintenance of fracture reduction according to radial height (Long plaster casts Vs Short plaster casts) | compared at baseline, at 7-10 days, at 4 weeks and at 12 weeks
  Radial height: distance between two parallel lines drawn perpendicular to the long axis of the radial shaft, one from the tip of the radial styloid and the other from the ulnar corner of the lunate fossa, normal 11-12 mm
To measure the maintenance of fracture reduction according to ulnar variance (Long plaster casts Vs Short plaster casts) | compared at baseline, at 7-10 days, at 4 weeks and at 12 weeks
  Ulnar variance: refers to the relative lengths of the distal articular surfaces of the radius and ulna, normal -4-+2 mm
To measure the maintenance of fracture reduction according to palmar tilt (Long plaster casts Vs Short plaster casts) | compared at baseline, at 7-10 days, at 4 weeks and at 12 weeks
  Palmar tilt: can be measured by obtaining the angle of intersection between a line drawn tangentially across the most distal points of the radial articular surface and a perpendicular to the midshaft of the radius, normal 0°-22°

SECONDARY OUTCOMES:
Correlation RX parameters Vs functional outcomes | twelve weeks
  To determine whether or not there is a direct correlation between radiological parameters and functional outcomes in conservatively treated patients for extra-articular distal radius fractures with dorsal displacement. The following will be used for the clinical evaluation: DASH, Mayo Wrist and Mayo Elbow scores.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Caruso, MD, Principal Investigator — Azienda Ospedaliero Universitaria di Ferrara
Locations (1):
- Azienda Ospedaliero Universitaria di Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caruso G, Tonon F, Gildone A, Andreotti M, Altavilla R, Valentini A, Valpiani G, Massari L. Below-elbow or above-elbow cast for conservative treatment of extra-articular distal radius fractures with dorsal displacement: a prospective randomized trial. J Orthop Surg Res. 2019 Dec 30;14(1):477. doi: 10.1186/s13018-019-1530-1. PMID 31888682